CLINICAL TRIAL: NCT07319871
Title: A Phase 1b Study of Pasritamig (JNJ-78278343), a T-cell Redirecting Agent Targeting Human Kallikrein 2 (KLK2), in Combination With JNJ-86974680, an A2a Receptor (A2aR) Antagonist, for Prostate Cancer
Brief Title: A Study of Pasritamig (JNJ-78278343) in Combination With JNJ-86974680 for Treatment of Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 78278343PBPCR1005; 78278343PBPCR1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Finding (Experimental): Participants will receive pasritamig in combination with JNJ-86974680 to determine the recommended phase 2 combination dose (RP2CD) regimen.
  Interventions: Drug: Pasritamig; Drug: JNJ-86974680
- Part 2: Dose Expansion (Experimental): Participants will receive pasritamig in combination with JNJ-86974680 at the RP2CD as determined in Part 1 of the study to confirm the safety and anti-tumor activity.
  Interventions: Drug: Pasritamig; Drug: JNJ-86974680

INTERVENTIONS:
Drug: Pasritamig — Pasritamig will be administered intravenously.
  Other Names: JNJ-78278343
Drug: JNJ-86974680 — JNJ-86974680 will be administered orally.

SUMMARY:
The purpose of this study is to identify the recommended phase 2 combination dose (RP2CD) of Pasritamig in combination with JNJ-86974680 in Part 1 (Dose finding) of the study and to determine how safe and tolerable the RP2CD is for treatment of participants with advanced prostate cancer in Part 2 (Dose expansion) of study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate. Primary small cell carcinoma, carcinoid tumor, neuroendocrine (NE) carcinoma, or large cell NE carcinoma arising in the prostate are not allowed; however, adenocarcinomas with NE features (for example [e.g.], immunohistochemistry [IHC] with both androgen receptor [AR]- and NE-marker positivity) are allowed
* Metastatic castration-resistant prostate cancer (mCRPC) that is metastatic either to bone, any lymph node, or both without clear evidence of metastasis to visceral organs. Local-regional invasion (rectum, bladder) and bone disease with soft tissue component can be included
* Prior orchiectomy or medical castration (for example, must be receiving ongoing androgen deprivation therapy with a gonadotropin-releasing hormone [GnRH] analog [agonist or antagonist] prior to the first dose of study drug and must continue this therapy throughout the treatment phase)
* Prostate-specific antigen (PSA) greater than or equal to (>=) 2 nanograms per milliliters (ng/mL) at screening
* Measurable or evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion criteria:

* Toxicity related to prior anticancer therapy that has not returned to grade less than or equal to (<=) 1 or baseline levels (except for alopecia, neuropathy [Grade 2] and vitiligo)
* Known allergies, hypersensitivity, or intolerance to any of the components (for example, excipients) of pasritamig or JNJ-86974680
* Active infection or condition that requires treatment with systemic antibiotics within 7 days prior to the first dose of study treatment. Antibiotic or antiviral prophylaxis is allowed
* Have leptomeningeal disease or brain metastases, except participants with definitively, locally treated brain metastases that are clinically stable and asymptomatic >2 weeks, and who are off corticosteroid treatment for at least 2 weeks prior to first dose of study treatment
* Any serious underlying medical conditions or other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site to understand the informed consent, or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-02-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) by Severity | Up to 1 year 2 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event. Cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines and ocular events will be graded using the alternative scale provided in the protocol.
Part 1: Number of Participants With Dose-Limiting Toxicity (DLT) | Up To Day 22
  High grade hematologic or non-hematologic toxicities with exceptions and/or toxicities leading to treatment discontinuation will be regarded as DLT.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 1 year 2 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the response evaluation criteria in solid tumors (RECIST) version 1.1 response criteria without evidence of bone progression according to prostate cancer working group 3 (PCWG3).
Prostate-Specific Antigen (PSA) Response Rate | Up to 1 year 2 months
  PSA response rate is defined as the percentage of participants with a decline of PSA of 50% or more from baseline.
Duration of Response (DOR) | Up to 1 year 2 months
  DOR will be calculated among responders (PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3 or RECIST version 1.1 response criteria, or death due to any cause, whichever occurs first.
Radiographic Progression-Free Survival (rPFS) | Up to 1 year 2 months
  rPFS is defined as the time from the date of first dose of pasritamig or JNJ-86974680 until the date of radiographic disease progression or death, whichever comes first.
Time to Response (TTR) | Up to 1 year 2 months
  TTR is defined for the responders as the time from the date of first dose of any study treatment to the date of first documented response.
Serum Concentration of Pasritamig | Up to 1 year 2 months
  Serum samples will be analyzed to determine concentrations of pasritamig.
Plasma Concentration of JNJ-86974680 | Up to 1 year 2 months
  Plasma samples will be analyzed to determine concentrations of JNJ-86974680.
Number of Participants With Anti-Pasritamig Antibodies | Up to 1 year 2 months
  Serum samples will be analyzed for the detection of anti-pasritamig antibodies using a validated assay method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Florida Cancer Specialists, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency